CLINICAL TRIAL: NCT02260011
Title: A Single-Dose, Double Blind, Crossover Trial to Determinate the Comparability of Ipratropium Bromide HFA-134a Inhalation Aerosol to the Market Standard, Atrovent® CFC Inhalation Aerosol, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study of the Comparability of Ipratropium Bromide Hydrofluoroalkane (HFA)-134a Inhalation Aerosol to the Market Standard, Atrovent® Chlorofluorocarbon (CFC) Inhalation Aerosol, in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 244.2498
Record Dates: First submitted 2014-09-11; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (5):
- Ipratropium bromide HFA-134a low (Experimental)
  Interventions: Drug: Ipratropium bromide HFA-134a inhalation aerosol
- Ipratropium bromide HFA-134a high (Experimental)
  Interventions: Drug: Ipratropium bromide HFA-134a inhalation aerosol
- Atrovent® CFC low (Active Comparator)
  Interventions: Drug: Atrovent® CFC inhalation aerosol
- Atrovent® CFC high (Active Comparator)
  Interventions: Drug: Atrovent® CFC inhalation aerosol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ipratropium bromide HFA-134a inhalation aerosol
  Arms: Ipratropium bromide HFA-134a high; Ipratropium bromide HFA-134a low
Drug: Atrovent® CFC inhalation aerosol
  Arms: Atrovent® CFC high; Atrovent® CFC low
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study was to compare the bronchodilator efficacy and safety of ipratropium bromide HFA-134a inhalation aerosol and marketed, Atrovent® CFC Inhalation Aerosol in COPD patients

ELIGIBILITY:
Inclusion Criteria:

All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

* Patients must have stable, moderate to severe airway obstruction with an FEV 1 (forced expiratory volume in the first second) <=65% of predicted normal and FEV1 <=70% of FVC (Forced Vital Capacity)

  * Males: Predicted normal FEV1=0.093 (height in inches) - 0.032(Age) - 1.343
  * Females: Predicted normal FEV1=0.085 (height in inches) - 0.025(Age) - 1.692
* Male or female patients 40 years of age or older
* Patients must have a smoking history of more than ten pack-years
* Patients must be able to demonstrate an improvement in FEV1 >=015% within one hour after inhalation of two puffs of Atrovent® inhalation aerosol (21 mcg per puff)
* Patients must be able to satisfactorily administer the medication, perform pulmonary function test and maintain records during the study period as required in the protocol
* All patients must sign an informed consent form prior to participation in the trial (i.e., prior to pre-study washout of their usual pulmonary medications and prior to fasting for laboratory tests)

Exclusion Criteria:

* Patients with significant disease other than COPD were will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with clinical relevant baseline hematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion, the patient is excluded
* All patients with serum glutamic oxaloacetic transaminase (SGOT) >80 IU/L; serum glutamic pyruvic transaminase (SGPT) >80 IU/L, bilirubin >2.0 mg/dL, or creatinine >2.0 mg/dL will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not to be conducted in these patients
* Patients with a history of asthma, allergic rhinitis or atopy or have a blood eosinophil count above 600/mm³. A repeat eosinophil count will not to be conducted in these patients
* Patients with a recent history (i.e., one year or less) of myocardial infarction
* Patients with a recent history (i.e., three years or less) of heart failure, patients with any cardiac arrhythmia requiring therapy, patients receiving any systemic beta blocker and patients on chronic daytime oxygen therapy
* Patients with known active tuberculosis
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed
* Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history or a thoracotomy for other reasons be evaluated as per exclusion criterion No. 1
* Patients with an upper respiratory tract infection or COPD exacerbation in the six weeks prior to screening visit (vist1) or during the baseline period
* Patients with known hypersensitivity to anticholinergic drugs
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients who are on cromolyn sodium or nedocromil sodium
* Patients who are on antihistamines
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g., oral contraceptives, intrauterine devices, diaphragm or Norplant®)
* Patients who have taken an investigational drug within one month or 6 half-lives (whichever is longer) of the drug prior to the screening visit or patients currently enrolled in other research study
* Patients with a history of and/or active alcohol or drug abuse

Exclusion criteria for patients with allergies

* Patients with active infectious rhinitis (common cold) as determined by history and physical
* Patients with upper or lower respiratory infection at screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2000-10; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) response, calculated as area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 6 (AUC0-6) | After each drug administration

SECONDARY OUTCOMES:
Changes in peak FEV1 response | Baseline and after each drug administration
Onset of therapeutic FEV1 response | After each drug administration
Duration of therapeutic FEV1 response | After each drug administration
Time to peak FEV1 response | After each drug administration
Forced Vital Capacity (FVC) AUC0-6 | After each drug administration
Changes from baseline in FEV1 | Baseline and after each drug administration
Number of patients with adverse events | Up to 5 month after first drug administration
Peak FVC response | After each drug administration
Changes from baseline in FVC | Baseline and after each drug administration